CLINICAL TRIAL: NCT04700215
Title: Comparison of Effectiveness of Bilevel Positive Airway Pressure and Incentive Spirometry in Reducing Post CABG Surgery Pulmonary Complications
Brief Title: Comparison of BiPAP and ٰIS in Reducing Post CABG Pulmonary Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaudhry Pervaiz Elahi Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, Muhammad Imran Khan, Doctor Muhammad Imran Khan, Chaudhry Pervaiz Elahi Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: No.01-2020/ED/CPEIC/MULTAN
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Complications
Keywords: CABG; BiPAP; IS
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 01 Effectiveness of BiPAP in reducing post CABG pulmonary complications (Active Comparator): Bilevel positive airway pressure device after every 6 hours
  Interventions: Device: BiPAP
- Group 02 Effectiveness of IS in reducing post CABG pulmonary complications (Active Comparator): Incentive spirometry for 15 minutes after every 4 hours
  Interventions: Device: Incentive spirometry

INTERVENTIONS:
Device: BiPAP — To give bilevel positive airway pressure to the lungs
  Other Names: Bilevel
  Arms: Group 01 Effectiveness of BiPAP in reducing post CABG pulmonary complications
Device: Incentive spirometry — IS for 15 minutes after every 4 hours
  Arms: Group 02 Effectiveness of IS in reducing post CABG pulmonary complications

SUMMARY:
To evaluate the effect of Bi-level Positive Airway Pressure (BiPAP) and Incentive Spirometry (IS) in post CABG patients.

DETAILED DESCRIPTION:
As postoperative pulmonary complications are major concern in cardiac surgery patients and our local data is deficient for making better management guidelines. My study aims to provide a base for future research on this dimension and to decide better management plan for post cardiac surgical pulmonary complications. The hypothesis is Post extubation BiPAP is more effective than Incentive Spirometry (IS) in reducing postoperative pulmonary complications in cardiac surgical patients and the purpose of the study is to evaluate the effect of Bi-level Positive Airway Pressure (BiPAP) and Incentive Spirometry (IS) in cardiac surgical patients.

This Randomized Controlled Trial (RCT) study will be conducted at Chaudhary pervaiz elahi institute of cardiology ICU multan.

A sample size of 350 patients will be taken and effect of BiPAP and Incentive spirometry will be studied in reducing pulmonary complications post CABG surgery. Data will be analyzed through SPSS. For quantitative variables, mean and standard deviation will be calculated and for qualitative variables, frequency and percentage will be calculated. Chi square test will be used to estimate association between qualitative variables. A p value < 0.05 will be significant.

ELIGIBILITY:
Inclusion Criteria:

* CABG patients
* Patient willing to study
* Patients planned for on-pump cardiac surgical procedures
* Both genders (Male & Female)
* Age 20-60 years
* Ejection fraction 40-60%

Exclusion Criteria:

* Patients with valvular lesions
* Off-pump cardiac surgery
* Refusal to give consent for BiPAP
* Emergency surgery
* Previous cardiac surgery
* Obesity BMI>30
* ASA status V

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Post CABG pulmonary complications | 06 months
  To see the effect of BiPAP and IS in reducing post CABG pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Imran Khan, MBBS, Principal Investigator — Chaudhry Pervaiz Elahi Institute of Cardiology
Locations (1):
- CPEIC, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No